CLINICAL TRIAL: NCT00966199
Title: Medication Induced Blood Pressure Reduction; Assessment of Cerebral Perfusion and Cognition in Hypertensive Elderly
Brief Title: The Effects of Blood Pressure Reduction on Cerebral Perfusion and Cognition in the Elderly Population
Acronym: MBRACE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Heart Foundation (Other)
Responsible Party: J.A.H.R. Claassen, MD, PhD, Radboud University Nijmegen Medical Centre
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MBRACE; 2008B113
Record Dates: First submitted 2009-08-17; First posted 2009-08-26 (Estimated); Last update posted 2009-08-26 (Estimated); Status verified 2009-08

CONDITIONS: Hypertension
Keywords: blood pressure; aging; cerebrovascular circulation; hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hypertensive elderly (Experimental): community dwelling hypertensive elderly from general practices
  Interventions: Drug: anti-hypertensive medication

INTERVENTIONS:
Drug: anti-hypertensive medication — 8-12 weeks of anti-hypertensive treatment with 2 weekly titration using registered hypertensive medication

SUMMARY:
The purpose of this study is to determine if a reduction in systolic blood pressure induced by anti-hypertensive medication results in changes in cerebral perfusion and cognition in hypertensive elderly. Hypertensive elderly will be treated using open-label anti-hypertensive medication for 8-12 weeks. Changes in cerebral perfusion and cognition will be assessed before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 70 years
* Systolic office blood pressure >= 160 mmHg
* Systolic home blood pressure >= 155 mmHg

Exclusion Criteria:

* Diabetes Mellitus
* Atrial fibrillation
* Dementia
* Renal failure requiring dialysis
* Life expectancy of less than 1 year
* Disabling stroke
* Contraindication for MRI or anti-hypertensive medication
* Systolic blood pressure > 220 mmHg

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-09; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Cerebral blood flow | T1, 8-12 weeks of treatment, T2

SECONDARY OUTCOMES:
Cognitive functioning assessed by neuropsychological testing | T1, 8-12 weeks of treatment, T2-3

CONTACTS AND LOCATIONS:
Overall Officials: Jurgen A Claassen, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University, Nijmegen, Gelderland, Netherlands